CLINICAL TRIAL: NCT04665583
Title: Single-Center, Prospective, Open-Label Study Standardizing a Prehabilitation Protocol to Optimize Patients Prior to Undergoing Tricuspid Intervention
Brief Title: Prehab Prior to Undergoing Tricuspid Intervention
Status: Terminated | Type: Observational
Why Stopped: Could not meet enrollment goal due to decrease in our target patient population (patients admitted for prehab).
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 020-101
Record Dates: First submitted 2020-11-23; First posted 2020-12-11 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Tricuspid Valve Disease; Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency | interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prehabilitation: All study patients will receive preoperative optimization with a standardized prehabilitation protocol prior to any intervention.
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — Prehabilitation will consist of careful pre-intervention assessment and personalized optimization, guided by Investigator judgment, with a specific focus on right ventricular function. This will be done by using a detailed echo acquisition protocol (Appendix 1). Assessments will be collected according to the schedule of events below (Table 1.). Therapy will include intravenous milrinone therapy and aggressive diuresis with evaluation for clinical and functional signs of improvement, according to standard of care.

SUMMARY:
This study will aim to standardize the prehabilitation protocol to optimize patients and document the clinical and echo variables that could improve clinical outcomes of tricuspid valve intervention.

DETAILED DESCRIPTION:
Prior to screening activities, each subject will be given an opportunity to ask questions and to understand the details of study participation. Subjects who meet the inclusion and exclusion criteria and have signed an informed consent form will be considered enrolled into the study. After a subject is consented and enrolled in the study, data will be collected prior to any intervention or surgery at the following time points: a) Screening/Baseline b) Day 1 of Prehab c) Day 2 of Prehab d) Day 3 of Prehab e) Day 4 of Prehab, f) and any data collected immediately prior to an intervention or incision (in the case of a surgical patient)

Subjects meeting eligibility criteria with planned tricuspid intervention will receive in-hospital optimization with THHBP's Prehab Protocol.

Prehabilitation will consist of careful pre-intervention assessment and personalized optimization, guided by Investigator judgment, with a specific focus on right ventricular function. This will be done by using a detailed echo acquisition protocol (Appendix 1). Assessments will be collected according to the schedule of events below (Table 1.). Therapy will include intravenous milrinone therapy and aggressive diuresis with evaluation for clinical and functional signs of improvement, according to standard of care. If there are clinical and functional signs of improvement before Day 4, and the subject is ready for TV surgery or any other intervention, they will have Day 4 procedures performed. After the tests and evaluations are completed, the Principal Investigator or Sub-Investigators will decide if the patient is a candidate for TV surgery or another intervention

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Moderate-Severe or Severe TR
3. Undergoing tricuspid valve surgical or catheter-based intervention

Exclusion Criteria:

1. Clinical instability according to the judgement of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 adult male or female patients undergoing tricuspid valve intervention at The Heart Hospital Baylor Plano
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Change in volume status according to daily input/outputs | 4-5 days (Day 1 to Day 4 of Prehab or day of surgical intervention)
  daily input/outputs (mL)
Change in volume status according to weight | 5-6 days (Baseline to Day 4 of Prehab or day of surgical intervention)
  daily weights (kg)
Change in Severity of Tricuspid Regurgitation by Echocardiographic assessment | 5 days (Baseline to Day 4 of Prehab)
  severity of tricuspid regurgitation (mild, moderate, severe)
Change in Nutritional Status | 4 days (Baseline to Day 3 of Prehab)
  Pre-albumin (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Heart Hospital - Plano, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We do not have a plan to shared IPD to researchers outside of our research team. We will make available aggregate data and results in the form of publications. Internal BSWH monitors will have access to IPD.

REFERENCES:
- [Background] Zack CJ, Fender EA, Chandrashekar P, Reddy YNV, Bennett CE, Stulak JM, Miller VM, Nishimura RA. National Trends and Outcomes in Isolated Tricuspid Valve Surgery. J Am Coll Cardiol. 2017 Dec 19;70(24):2953-2960. doi: 10.1016/j.jacc.2017.10.039. PMID 29241483
- [Background] Hamandi M, Smith RL, Ryan WH, Grayburn PA, Vasudevan A, George TJ, DiMaio JM, Hutcheson KA, Brinkman W, Szerlip M, Moore DO, Mack MJ. Outcomes of Isolated Tricuspid Valve Surgery Have Improved in the Modern Era. Ann Thorac Surg. 2019 Jul;108(1):11-15. doi: 10.1016/j.athoracsur.2019.03.004. Epub 2019 Apr 2. PMID 30951698
- [Background] Hamandi M, George TJ, Smith RL, Mack MJ. Current outcomes of tricuspid valve surgery. Prog Cardiovasc Dis. 2019 Nov-Dec;62(6):463-466. doi: 10.1016/j.pcad.2019.11.014. Epub 2019 Dec 2. PMID 31805294